CLINICAL TRIAL: NCT04402164
Title: Skeletally Versus Dentally Anchored Herbst Appliance During Treatment of Class 2 Mandibular Deficiency in Adolescent Patients; A CBCT Study
Brief Title: Skeletally Versus Dentally Anchored Herbst Appliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Salam Mohamed, Orthodontist, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlAzharU-189
Record Dates: First submitted 2018-01-29; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Angle Class II, Division 1
Keywords: Herbst, mini-plates, Skeletal Class 2 malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontic Appliances, Functional

STUDY DESIGN:
Intervention Model Description: Group 1: Dentally anchored Herbst appliance Group 2: Skeletally anchored Herbst appliance
Who Masked: Outcomes Assessor
Masking Description: another person than the investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dentally anchored Herbst group (Active Comparator): Herbst appliance will be anchored on the mandibular dentition
  Interventions: Device: Herbst appliance
- Skeletally anchored Herst group (Active Comparator): Herbst appliance will be anchored on mini-plates placed in the para symphesial areas
  Interventions: Device: Herbst appliance

INTERVENTIONS:
Device: Herbst appliance — telescopic appliance for mandibular advancement

SUMMARY:
The treatment of skeletal Class II malocclusion can be carried out through different approaches. One of these is the using of Fixed Functional Appliances (FFA), one of main drawbacks of these appliances is the proclination of the lower anterior teeth limiting the skeletal effect that is originally addressed in those patients.To overcome these limitations, miniplates anchored Forsus FRD were introduced, it showed high success rate in achieving a more skeletal effect with retroclination of lower anterior teeth rather than their proclination. Although Herbst appliance is categorized as the best FFA with more stable skeletal and dentoalveolar effects, miniplates had never been tried as an anchorage source with Herbst appliance in skeletal Class II patients.

DETAILED DESCRIPTION:
Skeletal Class II malocclusion is one of the most common orthodontic problems, which occurs in about one third of the population. Although there is many skeletal and dental combination that can contribute for the creation of Class II, however, mandibular retrusion is considered as the main contributing factor.

The treatment of skeletal Class II malocclusion can be carried out through three different time intervals. The first is an early treatment before the pubertal growth spurt through limiting the maxillary growth and stimulation of mandibular growth by using headgear and/or functional appliances. The second intervention would be during the maximum growth spurt through harnessing the spurt time to produce a more favorable skeletal effect by using of functional appliances either removable or fixed. Once growth had ceased, the third and last possible intervention would be one of the following treatment options; promoting the remaining growth through the usage of Fixed Functional Appliances (FFA), camouflage treatment and orthognathic surgery.

Fixed functional appliances (FFA) are aiming to stimulate mandibular growth by forward posturing the mandible to correct the skeletal antero-posterior discrepancy. Although there is always a controversy regarding the effectiveness of these appliances, many studies have been demonstrated successful correction of skeletal class II in adolescent patients through their use.

In a way to achieve this, it is recommended to use a rigid type of FFA like Herbst appliance and the Functional Mandibular Advancer rather than semi-rigid appliances like Forsus Fatigue Resistant Device (Forsus FRD).

Regardless of the patient's age, one of main drawbacks of these appliances is the proclination of the lower anterior teeth limiting the skeletal effect that is originally addressed in those patients.To overcome this limitation, mini screws had been used with both rigid and semi-rigid types of FFA. Incremental enhancement in the skeletal measurement has been noted by using them with the rigid type of FFA (e.g. Herbst appliance), however, the effect was still purely dentoalveolar when it came to semi rigid FFA (e.g. Forsus FRD), never to say that the success rate of these mini screws in the mandible is very low when compared with the maxilla which means a more complication and inconsistency in the clinical results.

To overcome these limitations, miniplates anchored Forsus FRD were introduced, it showed high success rate in achieving a more skeletal effect with retroclination of lower anterior teeth rather than their proclination. Although Herbst appliance is categorized as the best FFA with more stable skeletal and dentoalveolar effects,miniplates had never been tried as an anchorage source with Herbst appliance.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal Class II malocclusion due to mandibular deficiency (SNA=82+4, ANB ≥4o).
2. Overjet ≥5.0 mm.
3. All permanent dentition erupted with exception of the third molars.
4. The patient should be at the maturity stage of MP3-I (where the fusion of the epiphysis and metaphysis is completed according to the developmental stage of the middle phalanx).

Exclusion Criteria:

1. History of any medical problems that may interfere with orthodontic treatment.
2. Previous orthodontic treatment.
3. Clinical signs and symptoms of temporomandibular disorders.
4. Bad oral hygiene.

Ages: 14 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
condylar volume changes | 2 years
  volumetric changes that affects the condylar head when comparing pre and post treatment
amount of mandibular advancement | 2 years
  increase in mandibular length

SECONDARY OUTCOMES:
changes in inclination of lower anterior teeth | 2 years
  angular changes

CONTACTS AND LOCATIONS:
Overall Officials: Al-Dany A. Mohamed, Prof, Study Director — Al-Azhar University
Locations (1):
- AlAzharU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided